CLINICAL TRIAL: NCT01336608
Title: A 24-week Study to Evaluate the Effect of Fluticasone Furoate/Vilanterol 100/25 mcg Inhalation Powder Delivered Once-daily Via a Novel Dry Powder Inhaler on Arterial Stiffness Compared With Placebo and Vilanterol in Subjects With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: A 24-week Arterial Stiffness Study With Fluticasone Furoate/Vilanterol in COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113108
Record Dates: First submitted 2011-03-31; First posted 2011-04-18 (Estimated); Results first posted 2015-07-10 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Fluticasone Furoate/Vilanterol (Experimental): Inhaled corticosteroid/long acting beta-agonist
  Interventions: Drug: Fluticasone Furoate/Vilanterol
- vilanterol (Experimental): Inhaled long acting beta-agonist
  Interventions: Drug: Vilanterol
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone Furoate/Vilanterol — Inhaled corticosteroid/long acting beta-agonist
  Arms: Fluticasone Furoate/Vilanterol
Drug: Vilanterol — Inhaled long acting beta-agonist
  Arms: vilanterol
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
The purpose of the study is to investigate the effect of fluticasone furoate/vilanterol Inhalation Powder on arterial stiffness compared with placebo and vilanterol over a 24-week treatment period in subjects with COPD and aortic pulse wave velocity of 11.0 m/s or above.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis defined by ATS/ERS
* Former or current smoker
* A measured aortic pulse wave velocity = or > 11.0 m/s at Screening

Exclusion Criteria:

* Pregnancy
* A current diagnosis of asthma
* alpha1-antitrypsin deficiency as the underlying cause of COPD
* subjects with other and active respiratory disorders
* A cardiovascular event occurred in the 6 months prior to Visit 1
* Current severe heart failure (New York Heart Association Class IV) and have a known ejection fraction of < 30 %
* Clinical significant and uncontrolled hypertension
* Abnormal and clinical significant 12-lead ECG findings at Visit 1
* Have lung volume reduction or lung transplantation within 12 months prior to Visit 1
* Poorly controlled COPD: Acute worsening of COPD that is managed by subject with antibiotics or corticosteroids, or requires treatment prescribed by a physician in the 6 weeks prior to Visit 1; or subject needs to be hospitalised due to poorly controlled COPD within 12 weeks prior to Visit 1
* Lower respiratory tract infection that required use of antibiotics within 6 weeks prior to Visit 1
* Participate in the acute phase of a pulmonary rehabilitation within 4 weeks prior to Visit 1 or who will enter the acute phase of pulmonary rehabilitation during the study.
* Other diseases or abnormalities in the opinion of the investigator would put safety of the subject at risk through participation; or would affect the safety or efficacy analysis if the disease/condition exacerbated during the study.
* subjects with carcinoma has not been in complete remission for at least 5 years. Carcinoma in site of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded if the subject has been considered cured within 5 years since diagnosis.
* subjects with a history of hypersensitivity to any of the study medications or components of the inhalation powder.
* subjects with a known or suspected history of alcohol or drug abuse within the last 2 years prior to Screening
* subjects are medically unable to withhold albuterol or ipratropium for 4 hours prior to spirometry testing at each study visit
* subjects are medically unable to stop the 'excluded medications' listed in the protocol
* subjects started, discontinued certain medications listed in the protocol or have not been on a stable dose in the past three months prior to Screening, or are not anticipated to remain on a stable dose during the study treatment period.
* Long term oxygen therapy requiring >12 hour per day or a flow rate > 2 L/min
* A body mass index = or >35 kg/m2
* Fasting lipid level LDL>3.3 mmol/L, total cholesterol >5.2 mmol/L, and triglycerides > 2.24mmol/L
* Non-compliance
* Questionable validity of consent
* Prior use of study medication or other investigational drugs.
* Affiliation with investigator site

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2011-03-04 (Actual); Primary Completion 2014-11-04 (Actual); Study Completion 2014-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (65):
- United States (36):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Duluth, Georgia
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, Muncie, Indiana
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Traverse City, Michigan
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Fort Mill, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Edinburg, Texas
  - GSK Investigational Site, Abingdon, Virginia
- Germany (9):
  - GSK Investigational Site, Elsterwerda, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Norway (4):
  - GSK Investigational Site, Elverum
  - GSK Investigational Site, Kløfta
  - GSK Investigational Site, Moss
  - GSK Investigational Site, Stavanger
- Philippines (6):
  - GSK Investigational Site, Dagupan
  - GSK Investigational Site, Jaro, Iloilo City
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Marilao, Bulacan
  - GSK Investigational Site, Pasig
  - GSK Investigational Site, Quezon City
- South Korea (5):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Ilsanseo-gu, Goyang-si, Gyeonggi-do
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- Thailand (5):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Muang
  - GSK Investigational Site, Nan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113108 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113108 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113108 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113108 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113108 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113108 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113108 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 3011 participants (par.) were screened, 559 entered the Run-in Period (RIP), of whom 444 were randomized and received at least one dose of study medication; 430 of these were included in the Intent-to-Treat (ITT) Population.
Pre-assignment Details: Eligible par. at screening entered a 2-week, single-blind placebo RIP to obtain albuterol (salbutamol) use at Baseline, and to ensure that par.'s COPD was stable at randomization. At the end of the RIP, par. meeting the randomization criteria entered the double-blind treatment period (TP) of 24 weeks (Wk).
Groups:
- Placebo-Run-in: Participants received placebo once daily (QD) in the morning for 2 weeks. In addition, participants were provided an inhaled short-acting beta2-receptor agonist (SABA), albuterol (salbutamol) (metered dose inhaler [MDI] or nebules), to be used as a rescue medication for relief of chronic obstructive pulmonary disease (COPD) symptoms during the Run-in and Treatment Periods.
- Placebo QD: Participants received placebo QD in the morning via a dry powder inhaler (DPI) for 24 weeks. In addition, participants were provided an inhaled SABA, albuterol (salbutamol), to be used as a rescue medication for relief of COPD symptoms during the Run-in and Treatment Periods.
- VI 25 µg QD: Participants received vilanterol (VI) 25 micrograms (µg) inhalation QD in the morning via a DPI for 24 weeks. In addition, participants were provided an inhaled SABA, albuterol (salbutamol), to be used as a rescue medication for relief of COPD symptoms during the Run-in and Treatment Periods.
- FF/VI 100/25 µg QD: Participants received fluticasone furoate (FF)/VI 100/25 µg inhalation QD in the morning via a DPI for 24 weeks. In addition, participants were provided an inhaled SABA, albuterol (salbutamol), to be used as a rescue medication for relief of COPD symptoms during the Run-in and Treatment Periods.
Period: 2-week, Single-blind Run-In Period
Arm/Group | Placebo-Run-in | Placebo QD | VI 25 µg QD | FF/VI 100/25 µg QD
Started | 559 | 0 | 0 | 0
Completed | 444 | 0 | 0 | 0
Not Completed | 115 | 0 | 0 | 0
Not completed — Did Not Meet Continuation Criteria | 102 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Period: 24-week, Double-blind Treatment Period
Arm/Group | Placebo-Run-in | Placebo QD | VI 25 µg QD | FF/VI 100/25 µg QD
Started | 0 | 141 | 154 | 135
Completed the Treatment Period | 0 | 96 (Par. were considered to have completed the TP if they attended Visit 6 (Week 24).) | 124 (Par. were considered to have completed the TP if they attended Visit 6 (Week 24).) | 110 (Par. were considered to have completed the TP if they attended Visit 6 (Week 24).)
Completed | 0 | 97 (Par. completed study if attended Wk 24, had 1-wk follow-up contact and no early withdrawal.) | 124 (Par. completed study if attended Wk 24, had 1-wk follow-up contact and no early withdrawal.) | 111 (Par. completed study if attended Wk 24, had 1-wk follow-up contact and no early withdrawal.)
Not Completed | 0 | 44 | 30 | 24
Not completed — Adverse Event | 0 | 8 | 6 | 7
Not completed — Lack of Efficacy-No Sub-Reason | 0 | 2 | 0 | 0
Not completed — Lack of Efficacy-Sub-Reason Exacerbation | 0 | 13 | 13 | 6
Not completed — Protocol Violation | 0 | 4 | 3 | 3
Not completed — Protocol-defined Stopping Criteria | 0 | 4 | 3 | 6
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0
Not completed — Physician Decision | 0 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 7 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo QD: Participants received placebo QD in the morning via a DPI for 24 weeks. In addition, participants were provided an inhaled SABA, albuterol (salbutamol) , to be used as a rescue medication for relief of COPD symptoms during the Run-in and Treatment Periods.
- VI 25 µg QD: Participants received VI 25 µg inhalation QD in the morning via a DPI for 24 weeks. In addition, participants were provided an inhaled SABA, albuterol (salbutamol), to be used as a rescue medication for relief of COPD symptoms during the Run-in and Treatment Periods.
- FF/VI 100/25 µg QD: Participants received FF/VI 100/25 µg inhalation QD in the morning via a DPI for 24 weeks. In addition, participants were provided an inhaled SABA, albuterol (salbutamol) to be used as a rescue medication for relief of COPD symptoms during the Run-in and Treatment Periods.
- Total: Total of all reporting groups
Arm/Group | Placebo QD | VI 25 µg QD | FF/VI 100/25 µg QD | Total
Number analyzed (Participants) | 141 | 154 | 135 | 430
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.2 (8.10) | 68.7 (7.69) | 68.5 (8.01) | 68.5 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 36 | 31 | 89
  Male | 119 | 118 | 104 | 341
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 7 | 4 | 6 | 17
  Asian - Central/South Asian Heritage | 1 | 0 | 0 | 1
  Asian - East Asian Heritage | 21 | 23 | 18 | 62
  Asian - South East Asian Heritage | 45 | 51 | 47 | 143
  Asian - Mixed Race | 1 | 0 | 0 | 1
  White - Arabic/North African Heritage | 1 | 1 | 0 | 2
  White - White/Caucasian/European Heritage | 64 | 75 | 64 | 203
  Mixed Race | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (BL) in Aortic Pulse Wave Velocity (aPWV) at the End of the 24-week Treatment Period (Day 168)
Description: PWV is defined as the speed of travel of the pressure pulse along an arterial segment and can be obtained for any arterial segment accessible to palpation. aPWV is measured with tonometers positioned transcutaneously at the base of the common carotid artery and over the femoral artery. PWV increases with arterial stiffness and is defined by the Moens-Korteweg equation: PWV=square root of (Eh/2ρR), where E is Young's modulus of the arterial wall, h is the wall thickness, R is the arterial radius at the end of diastole, and ρ is the blood density. Change from BL was calculated as the Day 168 value minus the BL value. The analysis was performed using a repeated measures model with covariates of treatment, visit, age, gender, smoking history, history of exacerbation strata, geographical region, BL aPWV and interaction terms of BL by visit and treatment by visit.
Time Frame: BL to Day 168
Population: ITT Population: all randomized par. who received at least one dose of study medication. Number of par. presented represent those with data available at the time point being presented; however, all par. in the ITT population without missing covariate information and with at least one post BL measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: meters per second (m/sec)
Arm/Group | Placebo QD | VI 25 µg QD | FF/VI 100/25 µg QD
Number analyzed (Participants) | 85 | 117 | 103
meters per second (m/sec) | -1.97 (0.279) | -1.95 (0.241) | -1.75 (0.256)
Statistical Analysis 1: Comparison: Placebo QD vs VI 25 µg QD; Test type: Superiority or Other; p = 0.969, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least Squares Mean Difference = 0.01, 95% CI 2-sided [-0.71 to 0.74]
Statistical Analysis 2: Comparison: Placebo QD vs FF/VI 100/25 µg QD; Test type: Superiority or Other; p = 0.568, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least Squares Mean Difference = 0.22, 95% CI 2-sided [-0.53 to 0.96]
Statistical Analysis 3: Comparison: VI 25 µg QD vs FF/VI 100/25 µg QD; Test type: Superiority or Other; p = 0.566, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least Squares Mean Difference = 0.20, 95% CI 2-sided [-0.49 to 0.89]

2. Secondary Outcome: Change From BL in Clinic Visit Trough (Pre-bronchodilator and Pre-dose) FEV1 at Day 168
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled from the lungs in one second. Trough FEV1 measurements were taken electronically by spirometry at Screening, Days 1, 28, 84, 126, and 168. BL FEV1 was defined as the mean of the assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1. Trough FEV1 was defined as the mean of the FEV1 values obtained 24 hours after previous morning's dosing. Change from BL was calculated as the average at each visit minus the BL value. Analysis was preformed using a repeated measures model with covariates of visit, treatment, history of exacerbation strata, geographical region, BL FEV1 and interaction terms of BL by visit and treatment by visit.
Time Frame: BL to Day 168
Population: ITT Population. Number of par. presented represent those with data available at the time point being presented; however, all par. in the ITT population without missing covariate information and with at least one post BL measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | Placebo QD | VI 25 µg QD | FF/VI 100/25 µg QD
Number analyzed (Participants) | 96 | 123 | 111
Liters (L) | -0.049 (0.0221) | 0.033 (0.0202) | 0.106 (0.0210)
Statistical Analysis 1: Comparison: Placebo QD vs VI 25 µg QD; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.082, 95% CI 2-sided [0.023 to 0.141]
Statistical Analysis 2: Comparison: Placebo QD vs FF/VI 100/25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.155, 95% CI 2-sided [0.095 to 0.215]
Statistical Analysis 3: Comparison: VI 25 µg QD vs FF/VI 100/25 µg QD; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.074, 95% CI 2-sided [0.016 to 0.131]

3. Secondary Outcome: Mean Number of Occasions Rescue Medication [Albuterol (Salbutamol)] Used During a 24-hour Period Averaged Over the Entire 24-week Treatment Period
Description: Participants were given daily record cards for daily completion from BL (Week -1) through Week 24 (Visit 6) each morning and prior to taking study medication (i.e., single-blind and double-blind study medication) supplemental medication (albuterol [salbutamol] if received) and ipratropium bromide (if received). Participants recorded number of occasions supplemental albuterol/salbutamol (MDI and/or nebules) used over the previous 24 hours and any medical problems that they had experienced and any medication used to treat these medical problems over the previous 24 hours. Analysis was performed using an analysis of covarience (ANCOVA) model with covariates of treatment, BL mean of occasions of rescue medication use (Week -1), history of exacerbation, and geographical region.
Time Frame: BL (Week -1), Week 1 to Week 24
Population: ITT Population: all randomized participants who received at least one dose of study medication. Only those participants with at least 1 on treatment rescue medication measurement during the treatment period and without missing covariate information were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Occasions per 24 hours
Arm/Group | Placebo QD | VI 25 µg QD | FF/VI 100/25 µg QD
Number analyzed (Participants) | 139 | 152 | 135
Occasions per 24 hours | 1.97 (0.093) | 1.50 (0.089) | 1.47 (0.095)
Statistical Analysis 1: Comparison: Placebo QD vs VI 25 µg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Nominal p-value; Least Squares Mean Difference = -0.47, 95% CI 2-sided [-0.72 to -0.22]
Statistical Analysis 2: Comparison: Placebo QD vs FF/VI 100/25 µg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Nominal p-value; Least Squares Mean Difference = -0.50, 95% CI 2-sided [-0.76 to -0.24]
Statistical Analysis 3: Comparison: VI 25 µg QD vs FF/VI 100/25 µg QD; Test type: Superiority or Other; p = 0.803, ANCOVA; Least Squares Mean Difference = -0.03, 95% CI 2-sided [-0.29 to 0.22]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAE) and non-serious AEs were collected from the start of the double-blind (DB) treatment period (Visit 2) through the follow-up contact (7 days after Visit 6 [Week 25]).
Description: SAEs and non-serious AEs reported for par. of the Safety Population (Pop) comprised of ITT Pop plus par. from the excluded site who qualified for the ITT Pop. On-treatment AE or SAE is defined as an AE with an onset date on or after the start date of DB study medication, but not later than one day after the last dose of DB study medication.
Arm/Group | Placebo QD | VI 25 µg QD | FF/VI 100/25 µg QD
Serious Adverse Events (participants affected / at risk) | 5/145 | 12/158 | 9/141
Other Adverse Events (participants affected / at risk) | 24/145 | 27/158 | 34/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=145) | VI 25 µg QD (N=158) | FF/VI 100/25 µg QD (N=141)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways diseas (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 2
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=145) | VI 25 µg QD (N=158) | FF/VI 100/25 µg QD (N=141)
Nasopharyngitis (Infections and infestations) | 5 | 12 | 9
Oral candidiasis (Infections and infestations) | 1 | 2 | 9
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 4
Headache (Nervous system disorders) | 5 | 9 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.